CLINICAL TRIAL: NCT03896347
Title: A Randomized Study Evaluating ViBone®, Demineralized Bone Matrix, and Bone Morphogenetic Protein in 3-Level Oblique Lateral Lumbar Interbody Fusion
Brief Title: A Study Evaluating 3-Level OLIF Spine Fusion
Status: Withdrawn | Type: Observational
Why Stopped: Lack of enrollment
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-0003
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Spondylolisthesis; Retrolisthesis; Degenerative Disc Disease
Keywords: OLIF; ViBone; DBM; BMP; DDD
MeSH Terms: conditions — Spondylolisthesis; Intervertebral Disc Degeneration | interventions — Grafton demineralized bone matrix gel; Bone Morphogenetic Proteins

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- ViBone®: One product will be used on each level. At the time of surgery, implantation of ViBone®, DBM, and BMP will be randomized between the three treated levels.
  Interventions: Other: ViBone®; Other: Demineralized Bone Matrix; Other: Bone Morphogenetic Protein
- Demineralized Bone Matrix: One product will be used on each level. At the time of surgery, implantation of ViBone®, DBM, and BMP will be randomized between the three treated levels.
  Interventions: Other: ViBone®; Other: Demineralized Bone Matrix; Other: Bone Morphogenetic Protein
- Bone Morphogenetic Protein: One product will be used on each level. At the time of surgery, implantation of ViBone®, DBM, and BMP will be randomized between the three treated levels.
  Interventions: Other: ViBone®; Other: Demineralized Bone Matrix; Other: Bone Morphogenetic Protein

INTERVENTIONS:
Other: ViBone® — Viable bone allograft
Other: Demineralized Bone Matrix — Demineralized Bone Matrix
Other: Bone Morphogenetic Protein — Bone Morphogenetic Protein

SUMMARY:
The purpose of this study is to assess clinical and radiographic outcomes in patients who undergo three-level oblique lateral lumbar interbody fusion (OLIF) using ViBone, demineralized bone matrix (DBM), and bone morphogenetic protein (BMP). One product will be used on each level. Subjects will be followed for 12 months following surgery to assess degree of mineralization via computed tomography (CT) scan at 6 and 12 months, mean time to fusion, and maturation of fusion mass postoperatively via x-ray radiograph.

DETAILED DESCRIPTION:
Up to 120 patients undergoing three-level OLIF using ViBone, DBM, and BMP each on separate levels will be enrolled.

Implantation of ViBone, DBM, and BMP will be randomized between the three levels.

Subjects will be followed for a total of 12 months. Data and x-ray radiographs will be collected according to standard of care, including baseline, 3, 6, and 12 months post-surgery. Additionally, a CT scan will be required at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria

* Male or female, 18-80 years of age
* Patient must have degenerative disc disease, defined as discogenic back pain with degeneration of the disc confirmed by history and radiographic studies, affecting three contiguous levels between L2 and S1. Affected levels may also have up to Grade 1 spondylolisthesis or retrolisthesis
* Patient must have at least 6 months on non-operative treatment prior to study enrollment
* Patient signed Informed Consent Form
* Patient signed HIPAA Authorization (may be part of the ICF)
* Appropriate candidate for OLIF surgery using ViBone®, DBM, and BMP)
* Patient will adhere to the scheduled follow-up visits and requirements of the protocol
* Routine patient exams include pre-operative, operative, and three post-operative visits (3, 6, and 12 months post-surgery)
* CT scan of surgical site 6 and 12 months post-surgery

Exclusion Criteria

* Long-term, chronic use of medications that are known to inhibit fusion, bone metabolism, or immune suppressants 6 months prior to surgery (i.e., steroids, chemotherapy, DMARDs, etc.)
* Treatment with radiotherapy
* Patients who have who have had surgery for primary tumors or metastatic malignant tumors of the lumbar or sacral spine
* Nursing mothers or women who are pregnant or plan to become pregnant during the course of the study
* Current or recent history of malignancy or infectious disease. Patients with current or recent history of basal cell carcinoma are eligible.
* Inability to provide informed consent
* Rapid joint disease, bone absorption, osteomalacia, and/or diagnosed osteoporosis (bone density test score of <-2.5).
* Other medical or surgical conditions which would preclude the potential benefit of surgery, such as congenital abnormalities, immunosuppressive disease, elevation of sedimentation rate unexplained by other diseases, elevation of white blood count (WBC), or marked left shift in the WBC differential count.
* Morbid obesity as defined by a body mass index (BMI) of 40 or greater
* Patients with an allergy to titanium or titanium alloy
* Patients who are skeletally immature (<18 years of age or no radiographic evidence of epiphyseal closure)
* Active local or systemic infection or is undergoing adjunctive treatment for local or systemic infection.
* Patients with a known hypersensitivity to recombinant Bone Morphogenetic Protein-2, bovine Type I collagen, or to other components of the formulation of the BMP

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 120 male and female OLIF patients at up to 5 centers in the United States will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-13 (Actual)

PRIMARY OUTCOMES:
Graft Mineralization/Fusion | 12 months
  Degree of graft mineralization/fusion for each product via CT scan
Graft Mineralization/Fusion | 6 months
  Degree of graft mineralization/fusion for each product via CT scan

SECONDARY OUTCOMES:
Fusion Rates | 3, 6, and 12 months
  Fusion rates for each product as evidenced by bridging bone via x-ray radiograph
Time to Fusion | 3, 6, and 12 months
  Time to fusion for each product as evidenced by bridging bone via x-ray radiograph

OTHER OUTCOMES:
Complications and serious adverse reactions | Through study completion at 12 months
  Number of participants with ViBone®, DBM, or BMP-related complications and serious adverse reactions

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Sponsor website — http://www.aziyo.com